CLINICAL TRIAL: NCT06646562
Title: Long Acting Cabotegravir Plus Rilpivirine in People Living with HIV-1 Aged ≥ 60 Years for 24 Months.
Acronym: LOVER60
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMIB-LOVER60-2022-03; 2022-502882-53-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-11; First posted 2024-10-17 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: HIV-1 Infected Adults with Controlled Viremia

STUDY DESIGN:
Intervention Model Description: Phase IV study, prospective, open-label, single arm, multicentre, with a follow-up of 24 months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CAB LA + RPV LA (Experimental): the proportion of participants ≥60 years on stable oral ART that switch to CAB LA + RPV LA with plasma HIV-1 RNA ≥50 copies/mL at month 12 in the intention-to- treat exposed (ITT-E) population
  Interventions: Drug: Cabotegravir LA + Rilpivirine LA

INTERVENTIONS:
Drug: Cabotegravir LA + Rilpivirine LA — Cabotegravir (CAB) LA 600mg and Rilpivirine (RPV) LA 900mg will be administered intramuscularly every 2 months after an induction phase with a single administration in months 1 and 2.

SUMMARY:
People Living with HIV-1 (PLHIV) are an important group of patients attending their specialist's and continue growing thanks to efficacy antiretroviral treatment (ART), allowing them to stabilize the HIV-infection and to live a normal life despite the infection. The present study is encouraged to demonstrate that efficacy and security of CAB LA + RPV LA treatment's on this population remains the same compared to younger population of patients. This study also registers some metabolic and hepatic parameters to observe a hypothetical improvement on these parameters, as the population may suffer more comorbidities than younger population and therefore tolerability and convenience gains a huge importance on them. Psychosocial aspects are also very important in these patients as these patients may suffer social stigma, and therefore suffering certain psychological disorders.

ELIGIBILITY:
Inclusion Criteria:

* Be able to understand and comply with protocol requirements, instructions, and restrictions.
* Understand the long-term commitment to the study and be likely to complete the study as planned.
* Be considered appropriate candidates for participation in an investigative clinical trial with oral and intramuscularly injectable medications (e.g., no active substance use disorder, acute major organ disease, or planned long-term work assignments out of the country, etc.).
* Must be on a stable antiretroviral regimen without present or past evidence of viral resistance to, and no prior virological failure with agents of the NNRTI and INI class.
* Plasma HIV-1 RNA <50 copies/mL at screening.
* A female subject is eligible to participate if she is not pregnant (as confirmed by a negative serum hCG test at screen and a negative urine hCG test at randomization) and not lactating

Exclusion Criteria:

* Plasma HIV-1 RNA measurement ≥50 copies/mL within 6 months prior to screening. Blips are allowed (increased viral load ≥50 copies/mL but <200 copies/mL preceded and followed by a viral load less than 50 copies/mL)
* Any drug holiday during the window between initiating first HIV ART and 6 months prior to screening, except for brief periods (less than 1 month) where all ART was stopped due to tolerability and/or safety concerns.
* Any switch to a second line regimen, defined as change of a single drug or multiple drugs simultaneously, due to virologic failure to NNRTI or INSTI (defined as a confirmed plasma HIV-1 RNA measurement ≥200 copies/mL after initial suppression to <50 copies/mL while on first line HIV therapy regimen)
* Subjects who are currently participating in or anticipate being selected for any other interventional study. Observational studies and intervention studies that do not include treatments are allowed unless they interfere with scheduled visits.
* Participants receiving any prohibited medication and who are unwilling or unable to switch to an alternative medication

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Numer of patients on stable oral ART that switch to CAB LA + RPV LA with plasma HIV-1 RNA ≥50 copies/mL | Up to 12 Months
  Proportion of participants ≥60 years on stable oral ART that switch to CAB LA + RPV LA with plasma HIV-1 RNA ≥50 copies/mL at month 12 in the intention-to-treat exposed (ITT-E) population, per the FDA Snapshot algorithm.

SECONDARY OUTCOMES:
Levels of HIV-1 RNA Copies | 6, 12 and 24 Months
  To evaluate other estimations of virological control and number of episodes of plasma HIV-1 RNA ≥50 copies/mL that do not meet the criteria for confirmed virological failure
Levels of HIV-1 RNA Copies (plasma HIV-1 RNA ≥200 copies/mL) | 12 and 24 Months
  To determine the proportion of participants experiencing confirmed virologic failure
Number of Participants with experienced CVF (confirmed virologic failure) | 6, 12 and 24 Months
  To asses treatment emergent genotypic and phenotypic resistance in participants experiencing CVF. Levels of hiv-1 RNA copies
To evaluate the immune effects of switching to CAB LA + RPV LA | 6, 12 and 24 Months
  Plasma levels of (CD4 and CD4/CD8),
Number of SAES/SUSAR in patients treated with CAB LA + RPV LA | 6, 12 and 24 Months
  evaluation of parameters ensuring efficacy and security of patients, Number of SAES/SUSAR

OTHER OUTCOMES:
CD4/CD8 ratio | 6, 12 and 24 Months
  To assess the change in CD4/CD8 ratio
HIV Status | 6, 12 and 24 Months
  Questionnaire status version (HIVTSQs),
HIV Treatment Satisfaction | 6, 12 and 24 Months
  Perception of injection questionnaire (PIN)

CONTACTS AND LOCATIONS:
Locations (8):
- Spain (8):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Marina Baixa, Villajoyosa, Alicante
  - Hospital General Universitario Santa Lucía, Cartagena, Murcia
  - Hospital Universitario Rafael Mendéz de Lorca, Lorca, Murcia
  - Hospital General Universitario Reina Sofia, Murcia, Murcia
  - Hospital General Universitario Morales Meseguer, Murcia, Murcia
  - Hospital Clinico Universitario Virgen de la Arrixaca Murcia, Murcia, Murcia
  - Hospital General Universitario Los Arcos del Mar Menor, Pozo-Aledo, Murcia

IPD SHARING:
Plan to Share IPD: No